CLINICAL TRIAL: NCT05281770
Title: Non-interventional Study of the Austrian Headache Society: Monoclonal CGRP Antibodies for Migraine Prevention a Nationwide Real Life Study
Brief Title: Monoclonal CGRP Antibodies for Migraine Prevention - a Nationwide Real Life Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Austrian Migraine Registry Collaboration (Network)
Collaborators: Medical University of Vienna (Other); Medical University Innsbruck (Other); Austrian Headache Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: EK Nr: 1122/2021
Record Dates: First submitted 2021-12-23; First posted 2022-03-16 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-03

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura; Chronic Migraine; Episodic Migraine
Keywords: Erenumab; Galcanezumab; Fremanezumab; CGRP-antibodies
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura | interventions — erenumab; fremanezumab; galcanezumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Erenumab: Patients will be treated with this drug within standard of care treatment
  Interventions: Drug: Erenumab
- Galcanezumab: Patients will be treated with this drug within standard of care treatment
  Interventions: Drug: Galcanezumab
- Fremanezumab: Patients will be treated with this drug within standard of care treatment
  Interventions: Drug: Fremanezumab

INTERVENTIONS:
Drug: Erenumab — treatment with erenumab as chosen by treating physician
  Groups: Erenumab
Drug: Fremanezumab — treatment with fremanezumab as chosen by treating physician
  Groups: Fremanezumab
Drug: Galcanezumab — treatment with galcanezumab as chosen by treating physician
  Groups: Galcanezumab

SUMMARY:
The present non-interventional study on migraine prevention with monoclonal CGRP antibodies adresses questions concering safety, swichting from one CGRP mab to another, efficacy on auras in the real world setting.

DETAILED DESCRIPTION:
Introduction:

Monoclonal antibodies against calcitonin gene-related peptide (CGRP) or its receptor (CGRP-R) are an effective option for the preventative treatment in episodic and chronic migraine. All monoclonal antibodies against CGRP or CGRP-R have been proven efficacious in all various treatment endpoints (i.e. reduction of MMDs, improvement in Quality of Life etc.) in randomized phase 3 trials and were therefore approved by FDA and EMA. However, real world clinical experience/data in "non-study" patients is lacking as is data on long-term efficacy, elderly or data on switchers between antibodies that cannot be derived out of previous trials.

Phase 3 and 4 studies have addressed issues of efficacy and safety in highly selected clinical study populations and so far no safety concerns have emerged. However, long-term data are limited to a maximum period of 5 years and have been acquired in selected study cohorts probably not reflecting a "real world" patient population. It is a main goal of the study to acquire data on safety and efficacy in a real world setting where patients will be less selected than in clinical studies in terms of accompanying diseases or comorbidities. Another knowledge gap concerns the optimal procedure when switching the patient from one anti-CGRP therapy to another or being paused (and re-initiated) after a first successful treatment period. With specific evidence lacking, it is frequently recommended to wait several half-lives before initiating the next anti-CGRP therapy. Another unresolved question is whether non-responders to CGRP ligand blockers may respond to CGRP-receptor blockers and vice versa. While efficacy of anti-CGRP therapies has been demonstrated for migraine with and without aura, possible effects on the migraine auras per se have not been reported.

Phase 4 studies (non-interventional studies) on treatment with anti-CGRP therapies are being conducted in several countries in Europe. These are, however, limited to one specific substance. The proposed project will allow collecting data on the use of erenumab, fremanezumab, and galcanezumab on a nation- wide basis up to 36 months in a real-life setting.

The following knowledge should emerge from the registry:

Anti-CGRP therapies can be safely used in a wide spectrum of migraine patients with comorbidities and accompanying diseases over a long time period. There will be evidence how patients can be switched from one CGRP antibody to another. There will be an evidence base to switch anti-CGRP-therapies from ligand- to receptor- blockers or vice versa. Additionally the question whether a mAB even if effective should be paused or not after 1 year of treatment and what effect this pause might have will be addressed subsequently.

Methods Collected data will be entered in an electronic platform provided by Health Austria (https://goeg.at/) which has long-term experience in conducting and maintaining nation-wide registries, e.g. the Austrian Stroke Registry.

Non interventional study - The decision for therapy with an anti-CGRP monoclonal antibody/ CGRP antagonist is made by the treating physician and is NOT part of the Study. The study was approved by the relevant ethics committees and registered at a platform of the Austrian Agency for Health an Nutrition Safety at https://forms.ages.at/nis/. All patients treated in the headache centers are keeping headache diaries on paper or in electronic form as a standard of care procedure. Prospective and retrospective data collection from electronic charts is possible. Data are collected during routine visits which are scheduled in 3 months intervals. Collected data will be entered in an electronic platform provided by Health Austria (https://goeg.at/) in an anonymized form.

Study funding: Scientific reports concerning fremanezumab will be provideded to TEVA Austria, reports on erenumab to Novartis Austria and on galcanezumab to Eli Lilly Austria, based on financial compensation agreements.

ELIGIBILITY:
Inclusion Criteria (all of the follwing)

* episodic or chronic migraine with or without aura
* erenumab, fremanezumab or galcanezumab is prescribed as a standard of care treatment by treating physician Eptinezumab may be included as soon as available in Austria.

Exclusion Criteria:

• Off label use of erenumab, fremanezumab or galcanezumab

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male or female adult patients of at least 18 years or older in whom CGRP mabs can be prescribed according to Austrian regulations. These include treatment failure or intolerability / contraindications of at least 3 prophylactic medications. Documentation of treatment in a headache diary on paper or in digital format.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Migraine days per month (= 4 weeks) from baseline to month 6 | 6 months
  Either of the following: (i) patient has treated headache with a triptan (ii) criteria C+ D for migraine without aura are fulfilled (iii) criteria B+C for migraine with aura are fulfilled

SECONDARY OUTCOMES:
Change in headache days per month (= 4 weeks) from baseline to month 6 | 6 months
  Any day with headache
Change in aura days per month (= 4 weeks) from baseline to month 6 | 6 months
  Any day with at least one migraine aura
Change in days with acute headache medication per month (= 4 weeks) from baseline to month 6 | 6 months
  Any days on which medication against migraine was taken by the patient
Change in days with triptans per month (= 4 weeks) from baseline to month 6 | 6 months
  Any days on which triptans medication were taken by the patient
Change in headache intensity from baseline to month 6 | 6 months
  Usual intensity of headche attacks on a numerical rating scale from 1 -10. Higher numbers indicate more severe headache attacks
Change in unpleasantness of aura from baseline to month 6 | 6 months
  Usual unpleasantness of aura on a numerical rating scale from 1 -10. Higher numbers indicate more unpleasantness.
Change in migraine duration from baseline to month 6 | 6 months
  Usual duration of migraine headache attack
Change in migraine aura duration from baseline to month 6 | 6 months
  Usual duration of migraine aura

OTHER OUTCOMES:
Subjective change in quality of life from baseline to month 6 | 6 months
  3 point scale: improved, unchanged, worse
Change in MIDAS (Migraine Diasability Assessment Questionnaire) scores from baseline to month 6 | 6 months
  Migraine Disability Assessment Questionnaire. A higher Score indicates more disability. mnimum = 0, maximum =270
Change in impact of headache from baseline to month 6 | 6 months
  Questionnaire. Higher scores indicate more impact of headache. Minmum= 36, maximum =38
Adverse events | Up to 36 months. Assessment every 3 months, may differ between study centers.
  Any treatment emergent adverse events, Causality according to FDA rating: unlikely, possible, probable
Serious adverse events | Up to 36 months. Assessment every 3 months, may differ between study centers. Baseline refers to the 4 weeks interval before treatment start
  Definiation and causality according to FDA

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Broessner, Prof, Principal Investigator — Medical University Innbruck
Locations (3):
- Austria (3):
  - Medical University Innsbruck, Innsbruck, Tyrol
  - Medizinische Universität Wien, Vienna, Vienna
  - Clinic Hietzing, Vienna